CLINICAL TRIAL: NCT02967939
Title: Phase III Clinical Trial to Evaluate the Antiviral Activity and Safety of DA-2802(Tenofovir Disoproxil Orotate) and Viread®(Tenofovir Disoproxil Fumarate) in Chronic Hepatitis B Patients
Brief Title: Efficacy and Safety of DA-2802 in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA2802_HB_III
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis B， Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DA-2802 (Experimental): DA-2802 319mg tablet qd
  Interventions: Drug: DA-2802
- Viread® (Active Comparator): Viread® 300mg tablet qd
  Interventions: Drug: Viread®

INTERVENTIONS:
Drug: DA-2802 — DA-2802 319mg tablet qd + placebo tablet matching to Viread® 300mg.
  Other Names: tenofovir disoproxil orotate
  Arms: DA-2802
Drug: Viread® — Viread® 300mg tablet qd + placebo tablet matching to DA-2802 319mg.
  Other Names: tenofovir disoproxil fumarate
  Arms: Viread®

SUMMARY:
A study demonstrates the non-inferiority of DA-2802 when compared with ㅍViread® in chronic hepatitis B patients

DETAILED DESCRIPTION:
1. DA-2802 319mg Group: Administration with DA-2802 319mg tablet qd and placebo tablet matching to Viread® 300mg for 0-48 weeks.
2. Viread® 300mg Group: Administration with Viread® 300mg tablet qd and placebo tablet matching to DA-2802 319mg for 0-48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis B aged 18 years or older
* Subjects who have evidence to demonstrate a history of chronic hepatitis B for at least six months from the time of screening visit
* Subjects who have HBsAg positive test at screening visit
* Subjects who did not receive the hepatitis B treatment, including interferon or pegylated interferon, within 24 weeks of starting the screening test
* Subjects with an ALT of 80 units or more and 10 times lower than the normal upper limit at the time of screening

Exclusion Criteria:

* Subjects infected with hepatitis C, hepatitis D or human immunodeficiency virus
* Subjects with creatinine clearance of less than 50 ml/min at the screening visit
* At the time of screening visit, alpha-fetoprotein level was higher than 50 ng/ml and related imaging test showed hepatocellular carcinoma
* Subjects with decompensated liver disease who meet the following criteria:

  1. Total bilirubin levels greater than 2.5 mg/dl
  2. Prothrombin time is at least 3 seconds longer than normal upper limit
  3. Serum albumin value less than 30 g/l
  4. Subjects with a history of ascites, jaundice, bleeding from varicose veins, hepatic encephalopathy, or other signs of liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Difference of HBV DNA level(log10) | Change from baseline at 48 weeks

SECONDARY OUTCOMES:
Percentage of subjects HBV DNA < 400 copies/ml | at 24 weeks, 48 weeks
Percentage of subjects who had normal ALT levels | at 24 week, 48 week
Percentage of subjects who experienced loss of HBeAg | at 24 week, 48 week

CONTACTS AND LOCATIONS:
Overall Officials: Jong eun Yeon, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HJ, Kim JH, Yeon JE, Seo YS, Jang JW, Cho YK, Jang BK, Han BH, Lee C, Lee JH, Yoon JH, Kim KM, Kim MY, Kim DY, Park NH, Cho EY, Lee JS, Lee JW, Kim IH, Song BC, Lee BS, Kwon OS. A Multi-Center, Double-Blind Randomized Controlled Phase III Clinical Trial to Evaluate the Antiviral Activity and Safety of DA-2802 (Tenofovir Disoproxil Orotate) and Viread (Tenofovir Disoproxil Fumarate) in Chronic Hepatitis B Patients. J Korean Med Sci. 2022 Mar 21;37(11):e92. doi: 10.3346/jkms.2022.37.e92. PMID 35315603